CLINICAL TRIAL: NCT02291965
Title: Optimizing Busulfan: Efficacy, Toxicity, and Pharmacometabolomics
Brief Title: Blood Samples to Identify Biomarkers of Busulfan
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to end of funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Washington (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 9117; RG1001078 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2014-11-04; First posted 2014-11-17 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma; Immunodeficiency; Myelodysplastic Syndrome
Keywords: hematopoietic cell transplant
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Immunologic Deficiency Syndromes; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples from metabolomic and/or pharmacokinetic analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific Aim 1: To determine whether endogenous metabolomics-based biomarkers obtained before IV BU administration can predict IV BU clearance.

Specific Aim 2: To characterize IV BU metabolism by metabolomics.

Specific Aim 3: To identify covariates influencing IV BU pharmacokinetics.

DETAILED DESCRIPTION:
The long-range goal of this work is to improve overall survival in hematopoietic stem cell transplant (HCT) recipients by personalizing their conditioning regimen and/or intravenous (IV) busulfan (BU) doses using metabolomics. BU is an essential part of the majority of HCT conditioning regimens, but has a narrow therapeutic index; low BU plasma exposure (caused by rapid clearance) is associated with an increased risk of rejection or relapse, while high BU plasma exposure is associated with an increased risk of hepatotoxicity. Although pharmacokinetic (PK)-based dosing to a target BU exposure is often conducted, relapse and toxicity continue to be problematic. Furthermore, shorter IV BU courses necessitate alternative methods to personalize IV BU. IV BU clearance, however, is not associated with polymorphisms of glutathione S-transferase (GST) A1 and GSTM1, the predominant GSTs in BU conjugation with glutathione. Therefore, investigators seek to test the working hypothesis that metabolomic signature, which provides novel insight into the in vivo cellular response and metabolite identification, is associated with IV BU clearance. Investigators will first determine if endogenous metabolomics-based biomarkers obtained before BU administration can predict IV BU clearance. Researchers will evaluate endogenous biomarkers using a targeted (glutathione pathway) and global analyses via liquid chromatography-mass spectroscopy. In addition, investigators seek to evaluate IV BU metabolism using metabolomics in parallel with gas chromatography-mass selective detection in patients receiving PK-based IV BU. Researchers will evaluate plasma concentrations of eight different metabolites, building upon their experience with tetrahydrothiophene (THT+). To complement this metabolomic work, investigators seek to validate covariates associated with IV BU PK, specifically age and body size, to mitigate a typical challenge for metabolomics research: the lack of understanding of potentially confounding factors. FHCRC has been a reference clinical laboratory for PK-based BU dosing since 1996 and thus, FHCRC researchers have the largest database of IV BU PK. Using population pharmacokinetic (popPK) analysis, investigators will validate covariates for IV BU PK to guide future metabolomic studies. This popPK analysis can immediately improve patient care by using covariates to more accurately estimate an IV BU starting dose (i.e., before PK-based dosing) and by creating a limited sampling schedule to more efficiently use PK-based dosing. These complementary aims, which seek to identify novel metabolomics-based biomarkers, could overcome a critical barrier to HCT conditioning of balancing between response and toxicity. Based on compelling preliminary data, researchers expect to identify an endogenous metabolomic signature that will influence the choice of an IV BU starting dose with the intention of improving overall survival for patients receiving IV BU-containing HCT regimens.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive targeted intravenous busulfan (any dose, any number of doses, any dosing frequency) as part of their hematopoietic stem cell transplant conditioning;
* Weight > 21kg.

Exclusion Criteria:

* Unable to read English;
* Female patients who are pregnant or breastfeeding;
* Life expectancy severely limited by diseases other than malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving targeted IV busulfan as part of conditioning for a hematopoietic stem cell transplant
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Busulfan clearance | 24 hours after start of busulfan

SECONDARY OUTCOMES:
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine S. McCune, PharmD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States